CLINICAL TRIAL: NCT01475708
Title: Doxycycline in Therapy of Erythema Migrans - do the Accompanying Symptoms Influence the Outcome?
Brief Title: Doxycycline in Therapy of Erythema Migrans
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Franc Strle, M.D., PhD, University Medical Centre Ljubljana
Other Study IDs: EM-DOXY
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Lyme Borreliosis
Keywords: Lyme borreliosis; Erythema migrans; Doxycycline; Subjective symptoms; Outcome
MeSH Terms: conditions — Lyme Disease; Glossitis, Benign Migratory | interventions — Doxycycline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, cerebrospinal fluid, skin tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- no symptoms: patients with erythema migrans and no additional newly onset symptoms treated with doxycycline
  Interventions: Drug: Doxycycline
- mild symptoms: patients with erythema migrans and mild unspecific newly onset symptoms treated with doxycycline
  Interventions: Drug: Doxycycline
- severe symptoms-lumbar puncture: patients with erythema migrans and newly onset intense "neurologic" symptoms with lumbar puncture performed, treated with doxycycline
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — 100 mg PO bid, 14 days
  Other Names: Doxy

SUMMARY:
The investigators will compare the outcome of three groups of erythema migrans patients treated with doxycycline: a group without any accompanying symptoms, with mild symptoms and with severe symptoms that require lumbar puncture.

DETAILED DESCRIPTION:
Patients with erythema migrans treated with doxycycline for two weeks will be followed-up for one year (at 2 weeks, 2, 6 and 12 months) clinically and also by filling in the questionnaire to assess the presence of certain symptoms. Also the control group of their friends or relatives without a history of Lyme borreliosis will be included. The presence of their (unspecific) symptoms will also be recorded by the questionnaire at the time of enrollment and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* presence of erythema migrans
* >15 years old
* informed consent

Exclusion Criteria:

* pregnancy
* lactation
* multiple erythema migrans
* already treated with antibiotic for this episode of Lyme borreliosis
* allergy to doxycycline
* treatment with drugs with known interactions with doxycycline
* cerebrospinal fluid pleocytosis

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with erythema migrans reffered to Lyme Borreliosis outpatient clinic of the University Medical Center Ljubljana, Slovenia, Department of Infectious Diseases.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-05; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Comparing of objective sequelae and post-treatment subjective symptoms in three groups of erythema migrans patients treated with doxycycline: with no accompanying symptoms, with mild and with severe symptoms at the beginning. | 1 year follow-up

SECONDARY OUTCOMES:
Comparison of subjective symptoms between erythema migrans patients treated with doxycycline and control subjects without a history of Lyme borreliosis. | 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD PhD, Study Chair — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided